CLINICAL TRIAL: NCT04034498
Title: A Multicenter, International, Follow-up Study to Monitor the Efficacy and Safety of the Occlutech® Perimembranous Ventricular Septal Defect (PmVSD) Occluder in Patients With Perimembranous Ventricular Septal Defects
Brief Title: A Multicenter, International, Follow-up Study to Monitor the Efficacy and Safety of the Occlutech® PmVSD Occluder in Patients With Perimembranous Ventricular Septal Defects
Status: Active, not recruiting | Type: Observational
Sponsor: Occlutech International AB (Industry)
Responsible Party: Sponsor
Other Study IDs: Occ2018-01
Record Dates: First submitted 2019-07-18; First posted 2019-07-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Perimembranous Ventricular Septal Defect

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this registry is to gain more insight on the clinical use of the Occlutech perimembranous VSD occluder.

ELIGIBILITY:
Inclusion Criteria:

Patients with haemodynamically significant perimembranous defects which are located in the ventricular septum

Exclusion Criteria:

Occlutech® PmVSD Occluder is contraindicated for the following:

* Patients with defects less than 2 mm aortic rim and/or interference with the aortic or atrioventricular valves
* Patients less than 10.0 kg
* Patients with sepsis (local or generalized)
* Patients with left ventricle to right atrial shunting
* Patients with right to left shunting through the defect
* Patients with PmVSD with an aneurysm and multiple shunts that could not be successfully closed with one device
* Patients with complex heart lesions such as tetralogy of fallot
* History of repeated pulmonary infection
* Any type of serious infection 1 month prior to procedure
* Malignancy where life expectancy is less than 3 years
* Demonstrated intracardiac thrombi on echocardiography
* Patients with allergy to anti-platelet or anticoagulant therapy
* Patients with allergy to nickel and/or titanium and/or nickel/titanium based materials
* Patients with intolerance to contrast agents
* Patients with active bacterial infections
* Patients with very small vessels which are not suitable for recommended delivery sheath sizes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There will be no pre-selection of patients for enrollment in this registry. The criteria provided in the Instructions For Use should be followed. The study cohort will thus consist of consecutively enrolled patients at the discretion of the treating physician
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-07-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To confirm the efficacy of Occlutech PmVSD in patients requiring transcatheter occlusion (closure) of perimembranous ventricular septal defects. | 1 year following implantation
  The primary efficacy endpoint is defined as successful implantation of the device with a proper closure of the pmVSD (defined as reduction in VSD shunt of more than one grade as assessed by TTE post implantation).
To confirm the safety of Occlutech PmVSD in patients requiring transcatheter occlusion (closure) of perimembranous ventricular septal defects. | 1 year following implantation
  The primary safety endpoint is defined as absence of Serious Adverse Device Effects (SADEs) including procedure-related death, procedure-related stroke, systemic embolism, severe hemolysis, complete heart block requiring pacemaker implantation or device explantation, new-onset of severe tricuspid regurgitation (TR), new onset of severe aortic regurgitation (AR), device embolization, severe right-left ventricular outflow obstruction (RVOTO-LVOTO), cardiac tamponade, infective endocarditis or vascular complications requiring surgery.

CONTACTS AND LOCATIONS:
Locations (8):
- Children Health Ireland, Dublin, Ireland
- Thailand (2):
  - Queen Sirikit National Institute of Child Health, Bangkok
  - Prince of Songkla University, Hat Yai
- Turkey (Türkiye) (4):
  - Osmangazi University Faculty of Medicine Hospital, Eskişehir
  - Gaziantep University Hospital, Gaziantep
  - Izmir University of Health Sciences Tepecik Training and Research Hospital, Izmir
  - Kocaeli University Research and Application Hospital, Kocaeli
- City Children Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No